CLINICAL TRIAL: NCT02817750
Title: Pharmacokinetics Study of Zolpidem Hemitartarate Orodispersible Tablet 3.5 mg Formulation, With Fasting and Postprandial Administration, in Male and Female Healthy Volunteers, Produced by Biolab Sanus Farmacêutica Ltda
Brief Title: Pharmacokinetics Study of Zolpidem Hemitartarate Orodispersible Tablet 3.5 mg Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: JPJ 16/16
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: volunteers; Pharmacokinetics
MeSH Terms: interventions — Postprandial Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zolpidem hemitartarate (fasting + post-prandial) (Experimental): zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting and zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial
  Interventions: Drug: zolpidem hemitartarate tablet 3.5 mg (fasting + post-prandial)
- zolpidem hemitartarate (post-prandial + fasting) (Experimental): zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial and zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting
  Interventions: Drug: zolpidem hemitartarate tablet 3.5 mg (post-prandial + fasting)

INTERVENTIONS:
Drug: zolpidem hemitartarate tablet 3.5 mg (fasting + post-prandial) — zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting and zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial
  Arms: zolpidem hemitartarate (fasting + post-prandial)
Drug: zolpidem hemitartarate tablet 3.5 mg (post-prandial + fasting) — zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial and zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting
  Arms: zolpidem hemitartarate (post-prandial + fasting)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of the new formulation of zolpidem hemitartarate orodispersible tablet 3.5 mg in male and female healthy volunteers.

DETAILED DESCRIPTION:
This is a phase I study of zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting and postprandial administration. Sample size is 28 volunteers, male and female, aged from 18 to 50 years old.

This is an open-label, randomized, crossover study. Each volunteer will be randomized to one of the following sequencies:

* Sequency 1: zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting (period 1) and zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial (period 2)
* Sequency 2: zolpidem hemitartarate orodispersible tablet 3.5 mg postprandial (period 1) and zolpidem hemitartarate orodispersible tablet 3.5 mg in fasting (period 2) Formulation will be administered in a single dose, orally in each period. The volunteers will be admitted in two different periods of 36 hours each, when investigational product will be administered and blood samples will be collected at pre-determined periods of time up to 24 hours for pharmacokinetics evaluation.

Primary objective is to evaluate the pharmacokinetics of the new formulation of zolpidem hemitartarate orodispersible tablet 3.5 mg in healthy volunteers. As a secondary objective, it will be evaluated if there is any pharmacokinetics difference between genders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged from 18 to 50 years old (women cannot be pregnant or in breastfeeding period and should be committed to use an effective contraceptive method during the study)
* Body mass index (BMI) greater than or equal to 18.5 and less than or equal to 29.9 kg/m2
* Good health conditions or without significant diseases, according to best medical judgment, according to medical history, blood pressure and heart rate measurements, pulse, temperature, physical examination, electrocardiogram (ECG) and complementary laboratory tests
* Ability to understand the nature and objectives of the trial, including risks and adverse events, willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by informed consent form signature.

Exclusion Criteria:

* Know hypersensitivity to the investigational product (Zolpidem) or chemically related compounds
* History or presence of hepatic or gastrointestinal diseases, or other condition that interferes with drug absorption, distribution, excretion or metabolism
* Maintenance therapy with any drugs, except oral contraceptives
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic, psychiatric, cardiologic or allergic diseases of any etiology , that requires pharmacological treatment or considered as clinically relevant by the investigator
* Electrocardiographic findings that at investigator discretion are not recommended for study participation
* Deviations on screening laboratory results that are considered as clinically relevant by the investigator
* Smoking
* Intake of more than five cups of coffee or tea per day
* History of abusive use of drugs and alcohol
* Use of regular medication two weeks prior to study enrollment or use of any medications one week prior to study enrollment
* Hospitalization for any reasons up to 8 weeks prior to start of first period of trial treatment
* Treatment within 3 months prior to the start of trial treatment, with any drug with known and well-established toxic potential to major organs
* Participation in any pharmacokinetics trial with more than 300 mL of blood draw or administration of any experimental drug within 12 months prior to trial treatment start
* Donation or loss of 450 mL or more of blood within 3 months prior to trial enrollment or donation of more than 1500 mL of blood within 12 months prior to the trial treatment start
* Positive result for the BHCG urine test, performed by female subjects
* Positive results for the detection of abusive drugs at urine exam
* Result higher than 0.1 mg/L for the etilometer exam
* Any condition, according to investigator's best judgment, that prevents the subject to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve (0-last) | 24 hours
Area under the curve (0-inf) | 24 hours
Half life (t1/2) | 24 hours
Elimination rate constant (Ke) | 24 hours
Maximum serum concentration (Cmax) | 24 hours
Time to reach maximum (peak) plasma concentration following drug administration (tmax) | 24 hours
Volume of distribution (Vd) | 24 hours
Clearance (C) | 24 hours

SECONDARY OUTCOMES:
Number of adverse events | 60 days
Intensity of adverse events | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: José Pedrazzoli Júnior, PhD, Principal Investigator — UNIFAG - Universidade Integrada de Farmacologia e Gastroenterologia
Locations (1):
- UNIFAG - Unidade Integrada de Farmacologia e Gastroenterologia, Bragança Paulista, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No